CLINICAL TRIAL: NCT01228305
Title: Does Preoperative Acetaminophen Reduce Biochemical Markers of Oxidative Stress From Cardiopulmonary Bypass?
Brief Title: Acetaminophen for Oxidative Stress After Cardiopulmonary Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 090497
Record Dates: First submitted 2010-10-22; First posted 2010-10-26 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Congenital Heart Disease; Cardiopulmonary Bypass
Keywords: ventricular septal defect; atrioventricular septal defect; oxidative stress; cardiopulmonary bypass; acetaminophen; hemolysis; acute kidney injury; Congenital heart disease undergoing cardiopulmonary bypass
MeSH Terms: conditions — Heart Defects, Congenital; Heart Septal Defects, Ventricular; Atrioventricular Septal Defect; Hemolysis; Acute Kidney Injury | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acetaminophen (Experimental): Subjects will be randomly assigned to treatment using a permuted-block randomization algorithm. Acetaminophen will be given at a standard dose of 15 mg/kg IV every 6 hours for children >=2 years of age, 12.5mg/kg IV every 6 hours for children 29 days to <2 years of age, and 7.5mg/kg IV every 6 hours for neonates up to 28 days old for a total of 4 doses, starting shortly after intubation in the OR and before the start of CPB.
  Interventions: Other: Acetaminophen
- Placebo (Placebo Comparator): Subjects will be randomly assigned to treatment using a permuted-block randomization algorithm. Acetaminophen will be given at a standard dose of 15 mg/kg IV every 6 hours for children >=2 years of age, 12.5mg/kg IV every 6 hours for children 29 days to <2 years of age, and 7.5mg/kg IV every 6 hours for neonates up to 28 days old for a total of 4 doses, starting shortly after intubation in the OR and before the start of CPB.
  Interventions: Other: Acetaminophen

INTERVENTIONS:
Other: Acetaminophen — Acetaminophen will be given at a standard dose of 15 mg/kg IV every 6 hours for children >=2 years of age, 12.5mg/kg IV every 6 hours for children 29 days to <2 years of age, and 7.5mg/kg IV every 6 hours for neonates up to 28 days old for a total of 4 doses, starting shortly after intubation in the OR and before the start of CPB.
  Other Names: Tylenol

SUMMARY:
The current proposal tests the central hypothesis that acetaminophen will attenuate the oxidative stress response associated with cardiopulmonary bypass (CPB)-induced hemolysis in children undergoing cardiac surgery.

DETAILED DESCRIPTION:
Infants with complex congenital cardiac defects frequently undergo cardiopulmonary bypass (CBP) during surgical repair of their cardiac lesions (1). CBP exposes infants and children to endothelial damage, hyperoxia, hemolysis, and systemic inflammatory response (2-7). The systemic inflammatory response contributes to the organ dysfunction and is initiated by exposure of blood to the artificial surfaces of the extracorporeal circuit resulting in significant hemolysis and activation of complement. Hyperoxia has been shown to cause oxidative stress and the production of free radical molecules, which contributes to the morbidity of CPB. Hemolysis leads to free hemoglobin and the subsequent release of free iron in the plasma, which can catalyze redox reactions and has been shown to be another source of severe oxidant injury in children following bypass (8, 9). Additionally, the release of proinflammatory cytokines, hypothermia, hemorrhage requiring multiple transfusions, and activation of neutrophils leading to an enhancement of the respiratory burst contribute to oxidative injury and worsening inflammation (9).

Myoglobin and hemoglobin contain ferrous iron (Fe2+), which normally transports reversibly bound oxygen molecules to tissues. When muscle or red blood cells are damaged, the iron-chelating heme molecules are released into the plasma, and the ferrous iron is oxidized to the ferric (Fe3+) state. In the higher oxidation state, the ferric hemoproteins are able to reduce other molecules, notably hydrogen peroxide and lipid hydroperoxides, producing lipid peroxides and ferryl (Fe4+) hemoproteins. The ferryl hemoproteins can then enter an oxidation-reduction cycle with lipid molecules, causing further lipid peroxide production, leading to a cascade of oxidative damage to cellular membranes (10-12).

With increasing oxidative stress, oxygen free radicals attack esterified arachidonate layered within cell membrane lipid bilayers, resulting in the production of multiple lipid peroxidation products called isoprostanes (Iso-P) and isofurans (IsoF) (13-17). Many forms of IsoF and IsoP have been shown to be powerful vasoconstrictors, and have been shown to contribute to the pathogenesis and organ dysfunction associated with rhabdomyolysis, subarachnoid hemorrhage and hemolytic disorders (10, 16, 18-21). F2-isoprostanes are sensitive and specific markers of oxidative stress in vivo. (4) The mechanism/s causing increased oxidative stress during CPB are incompletely understood and the relationship between free hemoglobin and F2-isoprostanes in humans undergoing CPB is unknown.

Inhibition of hemoprotein-induced oxidative stress may have important clinical applications in humans. Hemolysis, in addition to contributing to the oxidative stress response, is also associated with acute kidney injury (AKI) in patients undergoing CPB or extracorporeal life support (5-6). In fact, plasma free hemoglobin has been shown to be an independent predictor of AKI in the early postoperative period (5). We have recently demonstrated that acetaminophen, through inhibition of prostaglandin H2-synthases (PGHS), inhibits the oxidation of free arachidonic acid catalyzed by myoglobin and hemoglobin. Moreover, in an animal model of rhabdomyolysis-induced kidney injury, acetaminophen significantly attenuated the decrease in creatinine clearance compared to control (10).

The current proposal tests the central hypothesis that acetaminophen will attenuate the oxidative stress response associated with CPB-induced hemolysis in children undergoing cardiac surgery. If acetaminophen attenuates the oxidative stress response associated with CPB-induced hemolysis the potential therapeutic benefit extends to all cardiac surgery patients requiring CPB. Based on the outcome of this pilot study we will design a prospective randomized trial to test the hypothesis that acetaminophen will reduce AKI associated with hemoprotein-induced oxidative stress following CPB.

ELIGIBILITY:
Patients will be eligible for enrollment based on the following inclusion criteria:

1) Infants or children (newborn to 17years of age) undergoing cardiopulmonary bypass for biventricular surgical correction of their congenital heart lesions.

Patients will not be eligible for this study based on the following exclusion criteria:

1. Patients scheduled for single ventricle palliation will be excluded, in an effort to standardize the time of repair, time on CPB, and surgical procedure.
2. Patients with severe neurological abnormalities at baseline.
3. Patients with major non-cardiac congenital malformations, developmental disorders or serious chronic disorders. Benign congenital malformations (such as club foot, ear tags, etc.) will not exclude the subject from the study.
4. Non-English speaking patients, or parent/legal guardians.
5. Patients less than 3 kg, to limit risk of excessive blood loss from lab draws.
6. Previous adverse reaction to acetaminophen
7. History of acute or chronic kidney disease
8. History of chronic liver disease
9. Emergency surgery

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2011-07; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
oxidative stress response as measured by F2-isoprostane | 24 hours after cardiopulmonary bypass
  Test the hypothesis that acetaminophen attenuates the oxidative stress response, as measured by F2-isoprostanes, in children undergoing cardiopulmonary bypass. The primary outcome is the oxidative stress response as measured by F2-isoprostane

SECONDARY OUTCOMES:
renal function | for the first 24 hrs after cardiopulmonary bypass
  Because free hemoglobin (hemolysis) has been associated with acute kidney injury (AKI) we will assess renal function as a secondary outcome in the immediate postoperative period. To assess renal function we will collect already available data including urine output, blood urea nitrogen, Creatinine and daily fluid ins and outs. Other potential confounders of AKI including cardiopulmonary bypass (CPB) time, daily use vasopressors and re-exploration for bleeding will be collected. In addition we will also measure urine neutrophil gelatinase-associated lipocalin (NGAL) as an early marker for AKI.

CONTACTS AND LOCATIONS:
Overall Officials: Scott A Simpson, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

REFERENCES:
- [Background] Allen BS, Ilbawi MN. Hypoxia, reoxygenation and the role of systemic leukodepletion in pediatric heart surgery. Perfusion. 2001 Mar;16 Suppl:19-29. doi: 10.1177/026765910101600i104. PMID 11334203
- [Background] Morita K, Ihnken K, Buckberg GD, Sherman MP, Young HH, Ignarro LJ. Role of controlled cardiac reoxygenation in reducing nitric oxide production and cardiac oxidant damage in cyanotic infantile hearts. J Clin Invest. 1994 Jun;93(6):2658-66. doi: 10.1172/JCI117279. PMID 8201004
- [Background] Haase M, Haase-Fielitz A, Bagshaw SM, Ronco C, Bellomo R. Cardiopulmonary bypass-associated acute kidney injury: a pigment nephropathy? Contrib Nephrol. 2007;156:340-53. doi: 10.1159/000102125. PMID 17464145
- [Background] Morrow JD. Quantification of isoprostanes as indices of oxidant stress and the risk of atherosclerosis in humans. Arterioscler Thromb Vasc Biol. 2005 Feb;25(2):279-86. doi: 10.1161/01.ATV.0000152605.64964.c0. Epub 2004 Dec 9. PMID 15591226
- [Background] Vermeulen Windsant IC, Snoeijs MG, Hanssen SJ, Altintas S, Heijmans JH, Koeppel TA, Schurink GW, Buurman WA, Jacobs MJ. Hemolysis is associated with acute kidney injury during major aortic surgery. Kidney Int. 2010 May;77(10):913-20. doi: 10.1038/ki.2010.24. Epub 2010 Feb 24. PMID 20182411
- [Background] Gbadegesin R, Zhao S, Charpie J, Brophy PD, Smoyer WE, Lin JJ. Significance of hemolysis on extracorporeal life support after cardiac surgery in children. Pediatr Nephrol. 2009 Mar;24(3):589-95. doi: 10.1007/s00467-008-1047-z. Epub 2008 Nov 12. PMID 19002722
- [Background] Kadiiska MB, Gladen BC, Baird DD, Germolec D, Graham LB, Parker CE, Nyska A, Wachsman JT, Ames BN, Basu S, Brot N, Fitzgerald GA, Floyd RA, George M, Heinecke JW, Hatch GE, Hensley K, Lawson JA, Marnett LJ, Morrow JD, Murray DM, Plastaras J, Roberts LJ 2nd, Rokach J, Shigenaga MK, Sohal RS, Sun J, Tice RR, Van Thiel DH, Wellner D, Walter PB, Tomer KB, Mason RP, Barrett JC. Biomarkers of oxidative stress study II: are oxidation products of lipids, proteins, and DNA markers of CCl4 poisoning? Free Radic Biol Med. 2005 Mar 15;38(6):698-710. doi: 10.1016/j.freeradbiomed.2004.09.017. PMID 15721980
- [Background] Christen S, Finckh B, Lykkesfeldt J, Gessler P, Frese-Schaper M, Nielsen P, Schmid ER, Schmitt B. Oxidative stress precedes peak systemic inflammatory response in pediatric patients undergoing cardiopulmonary bypass operation. Free Radic Biol Med. 2005 May 15;38(10):1323-32. doi: 10.1016/j.freeradbiomed.2005.01.016. PMID 15855050
- [Background] Laffey JG, Boylan JF, Cheng DC. The systemic inflammatory response to cardiac surgery: implications for the anesthesiologist. Anesthesiology. 2002 Jul;97(1):215-52. doi: 10.1097/00000542-200207000-00030. No abstract available. PMID 12131125
- [Background] Boutaud O, Moore KP, Reeder BJ, Harry D, Howie AJ, Wang S, Carney CK, Masterson TS, Amin T, Wright DW, Wilson MT, Oates JA, Roberts LJ 2nd. Acetaminophen inhibits hemoprotein-catalyzed lipid peroxidation and attenuates rhabdomyolysis-induced renal failure. Proc Natl Acad Sci U S A. 2010 Feb 9;107(6):2699-704. doi: 10.1073/pnas.0910174107. Epub 2010 Feb 1. PMID 20133658
- [Background] Ouellet M, Percival MD. Mechanism of acetaminophen inhibition of cyclooxygenase isoforms. Arch Biochem Biophys. 2001 Mar 15;387(2):273-80. doi: 10.1006/abbi.2000.2232. PMID 11370851
- [Background] Patel RP, Svistunenko DA, Darley-Usmar VM, Symons MC, Wilson MT. Redox cycling of human methaemoglobin by H2O2 yields persistent ferryl iron and protein based radicals. Free Radic Res. 1996 Aug;25(2):117-23. doi: 10.3109/10715769609149916. PMID 8885329
- [Background] Morrow JD, Hill KE, Burk RF, Nammour TM, Badr KF, Roberts LJ 2nd. A series of prostaglandin F2-like compounds are produced in vivo in humans by a non-cyclooxygenase, free radical-catalyzed mechanism. Proc Natl Acad Sci U S A. 1990 Dec;87(23):9383-7. doi: 10.1073/pnas.87.23.9383. PMID 2123555
- [Background] Montuschi P, Barnes PJ, Roberts LJ 2nd. Isoprostanes: markers and mediators of oxidative stress. FASEB J. 2004 Dec;18(15):1791-800. doi: 10.1096/fj.04-2330rev. PMID 15576482
- [Background] Milne GL, Musiek ES, Morrow JD. F2-isoprostanes as markers of oxidative stress in vivo: an overview. Biomarkers. 2005 Nov;10 Suppl 1:S10-23. doi: 10.1080/13547500500216546. PMID 16298907
- [Background] Roberts LJ 2nd, Fessel JP, Davies SS. The biochemistry of the isoprostane, neuroprostane, and isofuran Pathways of lipid peroxidation. Brain Pathol. 2005 Apr;15(2):143-8. doi: 10.1111/j.1750-3639.2005.tb00511.x. PMID 15912887
- [Background] Fessel JP, Porter NA, Moore KP, Sheller JR, Roberts LJ 2nd. Discovery of lipid peroxidation products formed in vivo with a substituted tetrahydrofuran ring (isofurans) that are favored by increased oxygen tension. Proc Natl Acad Sci U S A. 2002 Dec 24;99(26):16713-8. doi: 10.1073/pnas.252649099. Epub 2002 Dec 13. PMID 12482927
- [Background] Holt S, Moore K. Pathogenesis of renal failure in rhabdomyolysis: the role of myoglobin. Exp Nephrol. 2000 Mar-Apr;8(2):72-6. doi: 10.1159/000020651. PMID 10729745
- [Background] Holt S, Reeder B, Wilson M, Harvey S, Morrow JD, Roberts LJ 2nd, Moore K. Increased lipid peroxidation in patients with rhabdomyolysis. Lancet. 1999 Apr 10;353(9160):1241. doi: 10.1016/S0140-6736(98)05768-7. No abstract available. PMID 10217088
- [Background] Reeder BJ, Sharpe MA, Kay AD, Kerr M, Moore K, Wilson MT. Toxicity of myoglobin and haemoglobin: oxidative stress in patients with rhabdomyolysis and subarachnoid haemorrhage. Biochem Soc Trans. 2002 Aug;30(4):745-8. doi: 10.1042/bst0300745. PMID 12196184
- [Background] Roberts LJ 2nd. Inhibition of heme protein redox cycling: reduction of ferryl heme by iron chelators and the role of a novel through-protein electron transfer pathway. Free Radic Biol Med. 2008 Feb 1;44(3):257-60. doi: 10.1016/j.freeradbiomed.2007.10.042. Epub 2007 Dec 5. No abstract available. PMID 18067870